CLINICAL TRIAL: NCT00589407
Title: Unilateral Blindness/ Unilateral Deafness-relation to Neck Pain
Status: Terminated | Type: Observational
Why Stopped: there is a problem in recruting the paricipents
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Lemberg Hadas, Unilateral Blindness/ Unilateral Deafness-relation to Neck Pain, Hadassah Medical Organization
Other Study IDs: BARZ-001HMO-CTIL
Record Dates: First submitted 2007-12-23; First posted 2008-01-09 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Neck Pain; Unilateral Blindness; Unilateral Deafness
MeSH Terms: conditions — Neck Pain; Blindness; Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
Neck pain is a common complaint in the general population affecting 10-15% of the general population. females more than men. Known risk factors are: Trauma, Repetitive lifting of heavy objects at work, driving vibrating vehicles, frequents diving from boards and smoking. No study dealt with the possible role of unilateral loss of vision or hearing as a risk factor for the development of neck pain. Intuitively, one might suspect that unilateral blindness or deafness will lead to a tilted position of the head, in order to cover a better visual/audio field. This position, in time, might lead to the development of neck pain.

Our hypothesis is that patients with unilateral blindness/deafness will suffer from neck pain more frequently than the general population.

ELIGIBILITY:
Inclusion criteria:

* Men and women suffering from unilateral blindness or deafness
* Men and women visiting the ophthalmology or ENT clinics (general population) for reasons other than unilateral blindness/deafness and agreeing to participate in the study.
* Over 18 years of age
* Signed informed consent

Exclusion criteria:

* Subjects suffering from neck pain as a result of fractures, infection, or metastatic disease.
* Inability to understand or fill out the questionnaire/informed consent.

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: study group: patients with unilateral blindness and unilateral deafness as the control group: patients attending the eye ENT clinics for other reasons as control
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)

PRIMARY OUTCOMES:
neck pain | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yair Barzilay, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization., Jerusalem, Israel